CLINICAL TRIAL: NCT06423937
Title: A Single-center, Open-label, Double-cohort Clinical Study of Fruquintinib Plus Camrelizumab Plus HAIC in the Treatment of Non-MSI-H Advanced Colorectal Cancer Patients With Liver Metastasis After the Failure of First-line Treatment
Brief Title: Fruquintinib Plus Camrelizumab and HAIC in the Treatment of Non-MSI-H Advanced Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lu Wang, MD, PhD, Head of liver surgery department, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-SH-CRC-106
Record Dates: First submitted 2024-05-11; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advanced non-MSI-H left-sided colorectal cancer (Experimental): Advanced non-MSI-H left-sided colorectal cancer with liver metastasis after first-line standard treatment failure
  Interventions: Drug: combination therapy Combination: Fruquintinib plus Camrelizumab and HAIC (TOMOX/TOMIRI) Maintenance: Fruquintinib plus Camrelizumab
- Advanced non-MSI-H right-sided colorectal cancer (Experimental): Advanced non-MSI-H right-sided colorectal cancer with liver metastasis after first-line standard treatment failure
  Interventions: Drug: combination therapy Combination: Fruquintinib plus Camrelizumab and HAIC (TOMOX/TOMIRI) Maintenance: Fruquintinib plus Camrelizumab

INTERVENTIONS:
Drug: combination therapy Combination: Fruquintinib plus Camrelizumab and HAIC (TOMOX/TOMIRI) Maintenance: Fruquintinib plus Camrelizumab — Procedure/Surgery: HAIC After successful percutaneous hepatic artery cannulation, superior mesenteric arteriogram and hepatic arteriogram were performed, and after confirming that the subjects were eligible for enrollment according to the results, the hepatic artery was cannulated to the predetermined position. The catheter was connected to a syringe pump in the ward for continuous pumping of drugs.
  TOMOX（Raltitrexed 2 mg/m2, Oxaliplatin 85mg/m2）/ TOMIRI（Raltitrexed 2 mg/m2 ，Irinotecan 120mg/m2） Drug: Fruquintinib 3mg, qd, po, 21 days for a cycle, Suspend medication on the day of HAIC Drug: Camrelizumab 200mg, ivgtt,, 21 days for a cycle

SUMMARY:
Liver metastasis is the main cause of death in patients with colorectal cancer. The treatment of liver metastasis of colorectal cancer is the key to prolong the survival of patients. The purpose of this study was to investigate the efficacy and safety of fruquintinib combined with Camrelizumab and HAIC regimen in the treatment of non-MSI-H advanced colorectal cancer patients with liver metastasis after first-line standard treatment failure. Compared with the current standard second-line treatment plan, it provides new decisions for clinical practice, in order to reduce the adverse reactions of treatment and improve the tolerance and efficacy of patients. To provide more and more optimized medication options for patients with non-MSI-H advanced colorectal cancer complicated with liver metastasis.

DETAILED DESCRIPTION:
This is a single-center, open, double-cohort clinical study to explore the non-MSI-H type advanced colorectal cancer patients with liver metastases after the failure of first-line standard treatment with fruquintinib combined with calelizumab and HAIC.Clinically, systemic chemotherapy with 5-FU as the core, combined with irinotecan or oxaliplatin is the first-line and second-line standard chemotherapy regimen for unresectable CRLM patients, but various hepatotoxicity will occur during chemotherapy. HAIC can selectively deliver chemotherapeutic drugs to tumor cells, reduce hepatocyte toxicity, relatively preserve liver parenchyma, and increase the concentration of chemotherapy in the tumor. Tumor cells are exposed to chemotherapy for a longer time, which effectively improves the efficacy and safety of treatment. Anti-angiogenic drugs can hinder the growth of microvessels in tumors and the development of metastatic diseases. At present, multiple retrospective studies have provided evidence support. The response rate of HAIC combined with systemic targeted therapy can reach 74 % -92 %. Previous studies have suggested that anti-angiogenic drugs combined with immunotherapy is expected to be a treatment strategy for patients with advanced colorectal cancer who fail to receive standard treatment or cannot receive standard treatment. Therefore, this study investigated the efficacy and safety of fruquintinib combined with Camrelizumab and HAIC in the treatment of patients with non-MSI-H advanced colorectal cancer complicated with liver metastasis after first-line standard treatment failure.

ELIGIBILITY:
Inclusion Criteria:

* The subjects volunteered to join the study and signed informed consent, with good compliance and follow-up.
* Patients with histologically or cytologically confirmed non-MSI-H ( according to the detection criteria of the institutional testing center, immunohistochemistry, PCR or NGS detection can be used ) unresectable advanced colorectal cancer with liver metastasis ;
* Age ≥ 18 years, ≤75 years， male or female ;
* ECOG PS 0-1;
* Expected overall survival ≥3 months
* Patients must have at least one measurable liver metastases (RECIST 1.1)
* Patients who had only received one standard first-line systemic treatment and were confirmed to be ineffective, or could not tolerate first-line treatment ;
* Patients must have adequate organ and bone marrow function( No blood components and cell growth factors were used within 14 days before enrollment )
* Male or female patients with fertility voluntarily used effective contraceptive methods, such as double-barrier contraceptive methods, condoms, oral or injectable contraceptives, intrauterine devices, etc., during the study period and within 6 months of treatment in the last study. All female patients will be considered to have fertility, unless the female patient has natural menopause, artificial menopause or sterilization ( such as hysterectomy, bilateral adnexectomy or radioactive ovarian irradiation, etc. ), otherwise the female patient 's serum or urine test showed no pregnancy within 7 days before the study, and must be non-lactating patients.

Exclusion Criteria:

* Patients who are allergic or suspected to be allergic to the study drug or similar drugs
* Patients had other malignant tumors in the past 5 years or at the same time (except for the cured skin basal cell carcinoma and cervical carcinoma in situ);
* Participating in other clinical trials and received at least one treatment within 4 weeks before enrollment
* Patients with autoimmune disease or history of autoimmune disease within 4 weeks before enrollment
* patients currently have central nervous system (CNS) metastasis or previous brain metastasis and the symptom control time is less than 2 months
* Patients cannot take fruquintinib orally
* Patients who have received organ transplantation and bone marrow transplantation in the past
* Have taken other strong inducers or inhibitors of CYP3A4, P-gp substrates and BCRP substrates within 2 weeks before the First medication
* Received any operation (except biopsy) or invasive treatment or operation (except venous catheterization, puncture and drainage, etc.) within 4 weeks before enrollment
* Pleural effusion or ascites causing relevant clinical symptoms, including respiratory syndrome (dyspnea≥CTC AE grade 2)
* Clinically significant electrolyte abnormality#
* Systolic blood pressure > 140mmHg or diastolic blood pressure > 90mmHg regardless of any antihypertensive drugs; Or patients need more than two antihypertensive drugs
* Proteinuria ≥ 2+ (1.0g/24hr);
* Active gastric and duodenal ulcer, ulcerative colitis or uncontrolled hemorrhage in GI, or other conditions that may cause GI bleeding and perforation as determined by the investigator;
* Have evidence or history of bleeding tendency within 3 months or thromboembolic events within 12 months before enrollment( Hemorrhage > 30 mL within 3 months, hematemesis, black feces, hematochezia ), hemoptysis ( fresh blood > 5 mL within 4 weeks ) or thromboembolic events ( including stroke events and / or transient ischemic attack ) within 12 months ;
* Clinically significant cardiovascular disease, including but not limited to acute myocardial infarction, severe/unstable angina pectoris or coronary artery bypass grafting within 6 months before enrollment; NYHA classification > 2 Grade; ventricular arrhythmia requiring medical therapy; ECG showing QTc interval ≥ 480 ms
* Active or uncontrolled serious infection (≥CTCAE grade 2 infection)
* Pregnant or lactating women
* Any other disease, with clinically significant metabolic abnormalities, physical examination abnormalities or laboratory abnormalities, according to the judgment of investigator that the patient is not suitable for the the study drug (such as having epileptic seizures and require treatment), or would affect the interpretation of study results, or put patients at high risk
* Clinical uncontrolled active infections, including human immunodeficiency virus (HIV) infection, active hepatitis B / C (HBV DNA Positive[1×104 copies/mL or >2000 IU/ml], HCV RNA positive[>1×103 copies/mL]);
* Patients have other factors that may affect the results of the study or cause the study to be terminated halfway, such as alcoholism, drug abuse, other serious diseases (including mental diseases) that require concomitant treatment, and serious laboratory abnormalities. Accompanied by family or social factors, which will affect the safety of patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | 24 months
  Defined as percentage of participants achieving assessed complete response (CR) and partial response (PR) by the investigator according to the RECIST 1.1.

SECONDARY OUTCOMES:
disease control rate (DCR) | 24 months
  DCR was defined as the percentage of participants who have a confirmed complete response#CR# or partial response#PR# or stable disease#SD# per RECIST 1.1 as assessed by investigator
Progression-Free Survival (PFS) | 24 months
  PFS is defined as the time from enrollment to the first documented disease progression or death due to any cause, whichever occurs first. Responses are according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by investigator
Progression-Free Survival rate at 6 months | 6 months
  The proportion of patients who did not experience disease progression or death from treatment initiation to 6 months
overall survival (OS) | 24 months
  OS is the time from enrollment to death due to any cause.
Adverse events as assessed by NCI CTCAE v5.0 | 24 months
  overall incidence of adverse events (AE); incidence of grade 3 or higher AE; incidence of severe adverse events (SAE); incidence of AEs leading to discontinuation of drug use; incidence of AEs leading to suspension of drug use

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China